CLINICAL TRIAL: NCT00349076
Title: Prospective Randomised Multicenter Phase-III-study: Preoperative Radiochemotherapy and Adjuvant Chemotherapy With 5-Fluorouracil Plus Oxaliplatin Versus Preoperative Radiochemotherapy and Adjuvant Chemotherapy With 5-Fluorouracil for Locally Advanced Rectal Cancer
Brief Title: Neoadjuvant Chemoradiotherapy and Adjuvant Chemotherapy With 5-Fluorouracil and Oxaliplatin Versus 5-Fluorouracil Alone in Rectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAO/ARO/AIO-04; German Cancer Aid (no. 106759)
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms | interventions — Fluorouracil; Oxaliplatin

ARMS (2):
- 1 (Experimental): Preoperative simultaneous radiochemotherapy: 5-Fluorouracil und Oxaliplatin:
  Radiotherapy starts on day 1 of chemotherapy; 28 fractions; single dose: 1,8 Gy once per day, monday through friday; Total dose: 50,4 Gy; Oxaliplatin: 50 mg/m² i.v., days 1, 8, 22 und 29; 5-Fluorouracil: 250 mg/m²/d continuous infusion, days 1-14 and 22-35
  Adjuvant Chemotherapy:
  Oxaliplatin: 100 mg/m² i.v. on day 1; Calciumfolinate: 400 mg/m² on day 1; 5-Fluorouracil: 2400 mg/m² continuous infusion for 46 hours; repeat day 15, 8 cycles
  Interventions: Drug: 5-FU and oxaliplatin
- 2 (Active Comparator): Preoperative simultaneous radiochemotherapy: 5-Fluorouracil Radiotherapy starts on day 1 of chemotherapy; 28 fractions; single dose: 1,8 Gy once per day, monday through friday; Total dose: 50,4 Gy; 5-Fluorouracil: Days 1-5 and 29-33: 120h-continuous infusion 1000 mg/m²/d
  Adjuvant Chemotherapy: 5-Fluorouracil: 500 mg/m² on 5 consecutive days (day 1-5) i.v. bolus fot 2-5 minutes; repeat day 29, 4 cycles
  Interventions: Drug: 5-FU

INTERVENTIONS:
Drug: 5-FU and oxaliplatin — Preoperative radiochemotherapy:
  Oxaliplatin: 50 mg/m² i.v., days 1, 8, 22 und 29; 5-Fluorouracil: 250 mg/m²/d continuous infusion, days 1-14 and 22-35
  Adjuvant Chemotherapy:
  Oxaliplatin: 100 mg/m² i.v. on day 1; Calciumfolinate: 400 mg/m² on day 1; 5-Fluorouracil: 2400 mg/m² continuous infusion for 46 hours repeat day 15, 8 cycles
  Arms: 1
Drug: 5-FU — Preoperative radiochemotherapy:
  5-Fluorouracil: Days 1-5 and 29-33: 120h-continuous infusion 1000 mg/m²/d
  Adjuvant Chemotherapy: 5-Fluorouracil: 500 mg/m² on 5 consecutive days (day 1-5) i.v. bolus fot 2-5 minutes; repeat day 29, 4 cycles
  Arms: 2

SUMMARY:
Standard treatment for locally advanced cancer of the rectum is preoperative chemoradiotherapy with 5-Fluorouracil (5-FU) plus 4 cycles of postoperative chemotherapy with 5-FU. According to our previous study (CAO/ARO/AIO-94, published in the New England Journal of Medicine 2004; 351:1731-40) this treatment results in only 6% of local failures, yet, still 36% of all patients develop distant metastasis. Therefore, our new study (CAO/ARO/AIO-04) incorporates new drugs, i.e. 5-FU + oxaliplatin, in an effort to improve the control of distant metastases. It is our hypothesis that the rate of disease free survival will improve by 5 to 8% after 3 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age: 18 years
* Histologically proven, advanced primary carcinoma of the rectum (tumor ? 12cm from the anal verge, with clinically staged T3/4 or any node-positive disease
* No prior therapy except a diverting stoma
* ECOG PS less than or equal 2
* Adequate bone marrow function: Leukocytes > 3,5 x 10^9/L Absolute neutrophil count > 1,5 x 10^9/L Platelet count > 100 x 10^9/L Hemoglobin > 10 g/dl
* Adequate hepatic function: Total bilirubin < 2,0 mg/dl ALAT, ASAT, alkaline phosphatase, gamma-GT < 3 x ULN 7. Serum creatinine < 1,5 mg/dl, creatinine-clearance > 50 ml/min
* Written informed consent before randomization

Exclusion Criteria:

* Pregnant or breast feeding women
* Fertile patients without adequate contraception during therapy
* Past or ongoing drug abuse or alcoholic excess
* Prior chemotherapy
* Prior radiotherapy to the pelvis
* Prior (within 4 weeks) or concurrent treatment with any other investigational agent
* Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* History of severe somatic or psychological diseases: - instable cardiac disease not well controlled with medication, myocardial infarction within the last 6 months:* Central nervous system disorders or psychiatric disability including dementia or epileptic disease; * active uncontrolled intercurrent infections or sepsis
* Peripheral neuropathy > 2 (NCI CTC AE grading)
* Previous or concurrent malignancies, with the exception of adequately treated basal cell carcinoma of the skin or in situ carcinoma of the cervix. The inclusion of patients with other adequately treated tumors within the last 5 years has to be discussed with the principal investigator
* Chronic diarrhea (> NCI CTC AE-Grad 1)
* Known allergy to substances containing platinum compounds
* Concurrent use of the antiviral agent sorivudine or chemically related analogues
* Known deficiency of dehydropyrimidindehydrogenase (DPD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1256 (Actual)
Dates: Start 2006-07; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Disease free survival at 3 years defined as the interval from randomization to locoregional or metastatic recurrence or the appearance or a secondary colorectal cancer or death, whichever occurs first. | 3 years

SECONDARY OUTCOMES:
Resection rate, rate of sphincter preservation, tumor regression, cumulative incidence of local and distant recurrences, overall survival, toxicity, quality of life | 5-year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Sauer, M.D., Principal Investigator — Dept. of Radiation Therapy, University of Erlangen, Germany
Locations (89):
- Germany (89):
  - Kreiskliniken Altötting-Burghausen, Altötting
  - Gesundheitszentrum St. Marien, Amberg
  - Onkologische Gemeinschaftspraxis, Ansbach
  - Krankenhaus Marienwörth, Bad Kreuznach
  - Caritas-Krankenhaus, Bad Mergentheim
  - Onkologische Schwerpunktpraxis, Bad Soden
  - Klinik Bad Trissl-Oberaudorf, Bad Trissl
  - Klinikum Bayreuth GmbH, Bayreuth
  - Aerzteforum Hennigsdorf, Berlin
  - Städtische Kliniken, Bielefeld
  - St.-Agnes-Hospital Bocholt, Bocholt
  - St. Josef-Hospital, Bochum
  - Ruhr-Universität Bochum; Knappschaftskrankenhaus, Bochum
  - Klinikum Bremen-Mitte, Bremen
  - Onkologische Praxis, Buchholz
  - Praxis für Hämatologie und Onkologie, Burgwedel
  - Klinikum Coburg gGmbH, Coburg
  - Praxis für Hämatologie und Onkologie, Cologne
  - Gemeinschaftspraxis für Hämatologie und Internistische Onkologie, Cologne
  - Onkologisches Versorgungszentrum Rehling-Donauwörth-Dachau, Donauwörth
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Katholisches Krankenhaus St. Nepomuk, Erfurt
  - Dept. of Radiation Therapy, University of Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
  - Alfried Krupp Krankenhaus, Essen
  - Klinikum Esslingen a.N., Esslingen am Neckar
  - Universitätsklinikum, Frankfurt am Main
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Weisseritztal-Kliniken, Freital
  - Kliniken an der Paar, Krankenhaus Friedberg, Friedberg
  - Klinikum Fulda, Fulda
  - SRH-Waldklinikum, Gera
  - Wilhelm-Anton-Hospital, Goch
  - Klinik am Eichert, Göppingen
  - Georg-August-Universität Göttingen, Göttingen
  - Universitätsklinikum Greifswald, Greifswald
  - St. Elisabeth und St. Barbara Krankenhaus, Halle
  - Asklepios Klinik Hamburg-Harburg, Hamburg
  - Diakonie Klinikum Hamburg, Hamburg
  - Praxis für Hämatologie und Onkologie, Hamm, Hamm
  - Marienhospital, Herne
  - Onkologische Schwerpunktpraxis, Hildesheim
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Klinik für Knochenmarkstransplantation und Hämatologie/Onkologie GmbH, Idar-Oberstein
  - Klinikum der Friedrich Schiller Universität, Jena
  - Innere Medizin, Hämatologie und Int. Onkologie, Kassel
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Onkologische Schwerpunktpraxis, Kronach
  - Gemeinschaftspraxis Onkologie, Landshut
  - Klinikum Landshut, Landshut
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Universitätsklinikum - St. Hildegardis-Krankenhaus Mainz, Mainz
  - Phillips-Universität Marburg, Marburg
  - Kliniken Maria Hilf, Mönchengladbach
  - Gemeinschaftspraxis Onkologie, Muhr am See
  - Klinikum Schwäbisch Gmünd, Stauferklinik, Mutlangen
  - Universitätsklinikum Großhadern, München
  - Klinikum rechts der Isar, Technische Universität, München
  - Clemenshospital Münster, Münster
  - Universitätsklinikum Münster, Münster
  - Hämatologisch-onkologische Schwerpunktpraxis Northeim, Northeim
  - Klinikum Nürnberg, Nuremberg
  - Darmzentrum Ortenau, Offenburg
  - Klinikum Oldenburg; Pius Hospital Oldenburg, Oldenburg
  - Paracelsus-Krankenhaus Ruit, Ostfildern
  - St. Vincenz Krankenhaus, Paderborn
  - Klinikum Passau, Passau
  - St. Josefs Krankenhaus, Potsdam
  - Universitätsklinikum Regensburg, Regensburg
  - Schwerpunktpraxis für Hämatologie und Onkologie mit Tagesklinik, Regensburg
  - Krankenhaus Barmherzige Brüder, Regensburg
  - Klinikum Rosenheim, Rosenheim
  - Medizinische Fakultät der Universität Rostock, Rostock
  - Kreiskrankenhaus Rottweil, Rottweil
  - Thüringen-Kliniken Saalfeld-Rudolstadt, Saalfeld
  - Hämatologisch-Onkologische Schwerpunktpraxis, Singen
  - Onkologische Praxisgemeinschaft Stade, Stade
  - Klinikum Traunstein, Traunstein
  - Onkologische Schwerpunktpraxis Traunstein, Traunstein
  - Krankenhaus der Barmherzigen Brüder, Trier
  - Universitätsklinikum Ulm, Ulm
  - Marienhaus Klinikum, St. Elisabeth Klinik Saarlouis, St. Michael Krankenhaus Völklingen, Völklingen
  - Klinikum Wetzlar-Braunfels, Wetzlar
  - Asklepios Paulinen Klinik, Wiesbaden
  - Reinhard-Nieter-Krankenhaus, Wilhelmshaven
  - Juliusspital, Würzburg
  - Missionsärztliche Klinik, Würzburg
  - Universitätsklinikum Würzburg, Würzburg

REFERENCES:
- [Derived] Diefenhardt M, Fleischmann M, Martin D, Hofheinz RD, Piso P, Germer CT, Hambsch P, Grutzmann R, Kirste S, Schlenska-Lange A, Ghadimi M, Rodel C, Fokas E; German Rectal Cancer Study Group. Clinical outcome after total neoadjuvant treatment (CAO/ARO/AIO-12) versus intensified neoadjuvant and adjuvant treatment (CAO/ARO/AIO-04) a comparison between two multicenter randomized phase II/III trials. Radiother Oncol. 2023 Feb;179:109455. doi: 10.1016/j.radonc.2022.109455. Epub 2022 Dec 23. PMID 36572280
- [Derived] Diefenhardt M, Ludmir EB, Hofheinz RD, Ghadimi M, Minsky BD, Fleischmann M, Fokas E, Rodel C. Impact of body-mass index on treatment and outcome in locally advanced rectal cancer: A secondary, post-hoc analysis of the CAO/ARO/AIO-04 randomized phase III trial. Radiother Oncol. 2021 Nov;164:223-231. doi: 10.1016/j.radonc.2021.09.028. Epub 2021 Oct 4. PMID 34619239
- [Derived] Kosmala R, Fokas E, Flentje M, Sauer R, Liersch T, Graeven U, Fietkau R, Hohenberger W, Arnold D, Hofheinz RD, Ghadimi M, Strobel P, Staib L, Grabenbauer GG, Folprecht G, Kirste S, Uter W, Gall C, Rodel C, Polat B; of the German Rectal Cancer Study Group. Quality of life in rectal cancer patients with or without oxaliplatin in the randomised CAO/ARO/AIO-04 phase 3 trial. Eur J Cancer. 2021 Feb;144:281-290. doi: 10.1016/j.ejca.2020.11.029. Epub 2020 Dec 28. PMID 33383348
- [Derived] Diefenhardt M, Ludmir EB, Hofheinz RD, Ghadimi M, Minsky BD, Rodel C, Fokas E. Association of Treatment Adherence With Oncologic Outcomes for Patients With Rectal Cancer: A Post Hoc Analysis of the CAO/ARO/AIO-04 Phase 3 Randomized Clinical Trial. JAMA Oncol. 2020 Sep 1;6(9):1416-1421. doi: 10.1001/jamaoncol.2020.2394. PMID 32644104
- [Derived] Kitz J, Fokas E, Beissbarth T, Strobel P, Wittekind C, Hartmann A, Ruschoff J, Papadopoulos T, Rosler E, Ortloff-Kittredge P, Kania U, Schlitt H, Link KH, Bechstein W, Raab HR, Staib L, Germer CT, Liersch T, Sauer R, Rodel C, Ghadimi M, Hohenberger W; German Rectal Cancer Study Group. Association of Plane of Total Mesorectal Excision With Prognosis of Rectal Cancer: Secondary Analysis of the CAO/ARO/AIO-04 Phase 3 Randomized Clinical Trial. JAMA Surg. 2018 Aug 1;153(8):e181607. doi: 10.1001/jamasurg.2018.1607. Epub 2018 Aug 15. PMID 29874375
- [Derived] Hofheinz RD, Arnold D, Fokas E, Kaufmann M, Hothorn T, Folprecht G, Fietkau R, Hohenberger W, Ghadimi M, Liersch T, Grabenbauer GG, Sauer R, Rodel C, Graeven U; German Rectal Cancer Study Group. Impact of age on the efficacy of oxaliplatin in the preoperative chemoradiotherapy and adjuvant chemotherapy of rectal cancer: a post hoc analysis of the CAO/ARO/AIO-04 phase III trial. Ann Oncol. 2018 Aug 1;29(8):1793-1799. doi: 10.1093/annonc/mdy205. PMID 29873684
- [Derived] Rodel C, Graeven U, Fietkau R, Hohenberger W, Hothorn T, Arnold D, Hofheinz RD, Ghadimi M, Wolff HA, Lang-Welzenbach M, Raab HR, Wittekind C, Strobel P, Staib L, Wilhelm M, Grabenbauer GG, Hoffmanns H, Lindemann F, Schlenska-Lange A, Folprecht G, Sauer R, Liersch T; German Rectal Cancer Study Group. Oxaliplatin added to fluorouracil-based preoperative chemoradiotherapy and postoperative chemotherapy of locally advanced rectal cancer (the German CAO/ARO/AIO-04 study): final results of the multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2015 Aug;16(8):979-89. doi: 10.1016/S1470-2045(15)00159-X. Epub 2015 Jul 15. PMID 26189067
- [Derived] Rodel C, Liersch T, Becker H, Fietkau R, Hohenberger W, Hothorn T, Graeven U, Arnold D, Lang-Welzenbach M, Raab HR, Sulberg H, Wittekind C, Potapov S, Staib L, Hess C, Weigang-Kohler K, Grabenbauer GG, Hoffmanns H, Lindemann F, Schlenska-Lange A, Folprecht G, Sauer R; German Rectal Cancer Study Group. Preoperative chemoradiotherapy and postoperative chemotherapy with fluorouracil and oxaliplatin versus fluorouracil alone in locally advanced rectal cancer: initial results of the German CAO/ARO/AIO-04 randomised phase 3 trial. Lancet Oncol. 2012 Jul;13(7):679-87. doi: 10.1016/S1470-2045(12)70187-0. Epub 2012 May 23. PMID 22627104
- [Derived] Schirmer MA, Mergler CP, Rave-Frank M, Herrmann MK, Hennies S, Gaedcke J, Conradi LC, Jo P, Beissbarth T, Hess CF, Becker H, Ghadimi M, Brockmoller J, Christiansen H, Wolff HA. Acute toxicity of radiochemotherapy in rectal cancer patients: a risk particularly for carriers of the TGFB1 Pro25 variant. Int J Radiat Oncol Biol Phys. 2012 May 1;83(1):149-57. doi: 10.1016/j.ijrobp.2011.05.063. Epub 2011 Oct 12. PMID 22000747